CLINICAL TRIAL: NCT04980664
Title: Effort to Narrow the Gap Between in Accordance With Guidelines and Consent to Treat CHB Population in East of China
Acronym: GATE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Chao Wu, Principal Investigator, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IN-CN-320-6104
Record Dates: First submitted 2021-06-28; First posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Chronic Hepatitis b
Keywords: Chronic Hepatitis b; Antiviral treatment
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Integrated intervention strategies (Experimental)
  Interventions: Other: Integrated intervention strategies

INTERVENTIONS:
Other: Integrated intervention strategies — Implementation of integrated intervention strategies to reduce the proportion of indicated-but-not-treated CHB patients.

SUMMARY:
China has the world's largest burden of hepatitis B virus (HBV) infection and will be a major contributor towards the global elimination of hepatitis B disease by 2030. One of the main issues in the management of patients with chronic HBV infection (CHB) is to maximize the individuals who need the treatment engaged and retained in care. However, our investigation revealed that 21.1% patients were treatment eligible but not treated based on Chinese 2019 CHB treatment guidelines, while only 213 (13.9%) patients were indicated-but-not-treated according to AASLD 2018 Hepatitis B guidance in a real-life cohort study. To maximize the individuals who need the treatment engaged and retained in care, integrated intervention strategies to address these treatment barriers are urgently needed. Therefore, we aim to propose a study to narrow the gap between in accordance with guidelines and consent to treat CHB population in EAST of China.

ELIGIBILITY:
Inclusion Criteria:

1. Positive HBV surface antigen (HBsAg) for 6 months or more;
2. Elevated ALT levels (>1×ULN) and detectable HBV DNA;
3. Treatment-naïve;
4. Willing to attend this study and able to provide the written informed consent.

Exclusion Criteria:

1. Co-infection with other viral hepatitis and human immunodeficiency virus;
2. Concurrent with other chronic liver diseases, including primary biliary cirrhosis, autoimmune hepatitis, alcoholic hepatitis, nonalcoholic fatty hepatitis, and hereditary metabolic liver disease;
3. Patients with liver cirrhosis;
4. Coexistence of hepatocellular carcinoma and other malignant tumor;
5. Underwent liver transplantation before the enrollment;
6. Severe cardiac, renal, respiratory, hematological, or psychiatric illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of indicated-but-not-treated CHB patients. | 18 months
  The proportion of indicated-but-not-treated CHB patients.

SECONDARY OUTCOMES:
The proportion of lost to follow-up in CHB patients. | 18 months
The frequency of follow-up visit in CHB patients. | 18 months

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - The Third People's Hospital of Changzhou, Changzhou, Jiangsu
  - Huai'an No.4 People's Hospital, Huai'an, Jiangsu
  - Nanjing Drum Tower Hospital, The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - The Affiliated Infectious Diseases Hospital of Soochow University, Suzhou, Jiangsu